CLINICAL TRIAL: NCT03303417
Title: Effect of Kiwifruit on Gastrointestinal Fluid Distribution and Transit in Healthy Volunteers
Acronym: KIWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Zespri International Limited (Industry)
Responsible Party: Principal Investigator, Robin Spiller, Professor, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: A200317
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Constipation; Diet Modification
Keywords: Kiwifruit
MeSH Terms: conditions — Constipation | interventions — Magnetic Resonance Imaging; alcohol acyltransferase, Actinidia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: MRI analysis will be performed blind to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kiwifruit (Experimental): Participants asked to consume 2 kiwifruit twice a day for 3 days before undergoing MRI Scan
  Interventions: Diagnostic Test: MRI Scan; Other: Kiwifruit
- Control (Placebo Comparator): Participants asked to consume a calorie-matched sugar drink twice a day for 3 days before undergoing MRI Scan
  Interventions: Diagnostic Test: MRI Scan; Other: calorie-matched sugar drink

INTERVENTIONS:
Diagnostic Test: MRI Scan — Participants will undergo hourly MRI scans on day 3 to assess bowel fluid content
Other: Kiwifruit — Kiwifruit
  Arms: Kiwifruit
Other: calorie-matched sugar drink — calorie-matched sugar drink
  Arms: Control

SUMMARY:
Constipation is a widespread and common problem in which a person finds it difficult and/or painful to open their bowels. The current treatment is the use of medications called laxatives. Kiwifruit is a widely available food that has been shown to possess some laxative properties. The cause of this is unknown. Non-invasive medical imaging techniques such as Magnetic Resonance Imaging now allow taking pictures of the gut and its contents. The Nottingham GI MRI research group specialises in these techniques and in this study use such images to assess the changes induced in the gut contents by kiwifruit to improve understanding of how it helps patients with constipation.

The volunteers will be asked to undergo 2 studies in which they take either kiwifruit or placebo (sugary drink) two times a day for 2 days and then spend a study day where will they will be fed some more kiwifruit/placebo and some normal food and image their gut at intervals. Participants will be asked to complete a stool diary to determine if they experience a laxative effect.

DETAILED DESCRIPTION:
1. Background. Chronic constipation affects approximately 17% of the population worldwide and remains an important unmet need since patients are currently often dissatisfied with treatment Current treatments which stimulate propulsive colonic motility or osmotic laxatives are successful in increasing stool frequency but are often associated with bloating, cramps and abdominal discomfort. Furthermore, such powerful treatments taken intermittently often create abnormal colonic contents and may result in alternation between diarrhoea and no stools. Many patients would benefit from a less powerful treatment which could be taken daily. Kiwifruit offer such an alternative and have been shown to increase stool volume and frequency. The mode of action however is unclear. Kiwi is 3% fibre (approximately 1/3 insoluble) and contains around 3% nonstarch polysaccharide including pectins, hemicellulose and cellulose, with high water holding capacity 1.5 times that of ispaghula, a commonly used laxative. Using recently developed and validated novel non-invasive MRI techniques, the University can assess transit and fluid distribution in the small intestine [4]. The University has also developed methods to assess colonic fluid, volumes and motility.
2. Aims. To assess the effect of kiwifruit on gastrointestinal fluid distribution.
3. Experimental protocol and methods. A randomised, placebo controlled, 2-way cross-over study in N=15 healthy volunteers assessing the response (versus baseline values) of 2 kiwifruit b.d vs placebo (28 gm maltodextrin drink providing 120kcal equal to that of 2 kiwifruit) daily. After a screening visit to confirm eligibility, study subjects will be randomised as to the test product schedule. Subjects will complete a daily stool diary documenting stool frequency and consistency using the Bristol Stool Form Scale. They will consume the test product allocated starting on Day 4. At 9 am of the morning of Day 5 they will ingest 5 MRI transit markers as described below and note the time of ingestion. The markers will be imaged at 24 hours (baseline scan of Day 6). On the main study day, the subjects will arrive fasted overnight and undergo fasting scans before consuming that day's allocated test product with 250ml of water. After 30 minutes considered to be Time =0 they will consume a standard rice pudding meal as used in previous studies. They will then undergo serial scanning hourly for 7 hours taking the second dose of test product plus 250ml water at Time 180 minutes. The third dose is taken at 320 minutes followed at 380 minutes by a second, larger test meal consisting of 400 g microwaveable macaroni cheese ready meal (Sainsbury), 100 g cheesecake slice (Sainsbury), and 250 mL bottled still water. The second test meal provides approx. 1000 kcal. The final scan will at time 420 minutes to assess the effect of ileal emptying on gastrointestinal fluid distribution. They will then be allowed home. There will be 2 weeks between studies to ensure return to baseline. At the end of the study a further 3 participants will be scanned in exactly the same protocol however at a lower dose of kiwifruit (2 fruit once daily) to determine if the effect is still visible.
4. Measurable end points/statistical power of the study. Primary endpoint: Effect of Kiwifruit on Ascending colon T1 area under curve from time 0-420.

Secondary endpoints: Effect of Kiwifruit on the following measures both fasting and postprandial AUC 0-420 minutes: 1) small bowel water content 2) ascending (AC), transverse (TC) and descending (DC) colonic volumes. 3) Transit of markers through gut as assessed by the weighted position score at 24 h (WAPS24) 4) Colonic motility 5) Gastric emptying of test meal 6) T1 of AC and DC. Pilot data with a standard laxative dose of ispaghula 7g t.d.s. showed a change of T1 AUC 0-360 of mean (SD) 88 (55) sec.min . Using this data n=15 healthy volunteers will give us >90% power to detect such a difference.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers scoring within the normal range for bowel symptoms as assessed using the GSRS, aged 18-65 years.

Exclusion Criteria:

1. Inability to discontinue medication likely to alter GI transit.
2. Previous gastrointestinal surgery (excluding cholecystectomy and appendectomy).
3. Known inflammatory bowel disease, coeliac disease.
4. Known intolerance of kiwifruit.
5. Inability to discontinue drugs likely to alter gut transit.
6. Subjects considered by the investigator unlikely to comply with study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 healthy volunteers were recruited from the population of Nottingham and surroundings. 2 dropped out after a single visit due to unexpected work commitments so 14 volunteers completed the study
Groups:
- Kiwifruit Then Control: Participants asked to consume 2 kiwifruit twice a day for 3 days before undergoing MRI Scan MRI Scan: Participants will undergo hourly MRI scans on day 3 to assess bowel fluid content Kiwifruit: Kiwifruit.
  Washout period of 2 weeks
  Then
  Participants asked to consume a calorie-matched sugar drink twice a day for 3 days before undergoing MRI Scan MRI Scan: Participants will undergo hourly MRI scans on day 3 to assess bowel fluid content calorie-matched sugar drink: calorie-matched sugar drink
- Control Then Kiwifruit: Participants asked to consume a calorie-matched sugar drink twice a day for 3 days before undergoing MRI Scan
  MRI Scan: Participants will undergo hourly MRI scans on day 3 to assess bowel fluid content
  calorie-matched sugar drink: calorie-matched sugar drink
  Washout of 2 weeks
  Then Participants asked to consume 2 kiwifruit twice a day for 3 days before undergoing MRI Scan MRI Scan: Participants will undergo hourly MRI scans on day 3 to assess bowel fluid content Kiwifruit: Kiwifruit
Period: Overall Study
Arm/Group | Kiwifruit Then Control | Control Then Kiwifruit
Started | 8 | 8
Completed | 7 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: 14 participants completed the study
Groups:
- All Study Participants: All participants randomised to either "Kiwifruit then Control" or "Control then Kiwifruit" Interventions
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 26 [21 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 14
BMI [Mean (Full Range); unit: kg/m^2] | 23 [17.6 to 30.1]

OUTCOME MEASURES:

1. Primary Outcome: Relaxation Time in Ascending Colon
Description: Area under curve of Ascending colon T1 measured on MRI , in milliseconds. Measurements at 0, 1, 2, 3, 4, 5, 6, 7, and 8 hours post-intervention
Time Frame: 0 - 8 hours
Measure: Mean (Standard Deviation); unit: seconds*minutes
Arm/Group | Kiwifruit | Control
Number analyzed (Participants) | 14 | 14
seconds*minutes | 312 (92) | 256 (97)

2. Secondary Outcome: Small Bowel Water Content Measured by MRI, in mL
Description: Area under the curve of change of small bowel water, 0-8 hours, measured by MRI, in mL Measurements at 0, 1, 2, 3, 4, 5, 6, 7, and 8 hours post-intervention
Time Frame: 0 - 8 hours
Population: 14 participants completed the study
Measure: Mean (Standard Deviation); unit: ml*minutes
Arm/Group | Kiwifruit | Control
Number analyzed (Participants) | 14 | 14
ml*minutes | 85530 (34923) | 35023 (15557)

3. Secondary Outcome: Colonic Volume
Description: Ascending (AC), transverse (TC) and descending (DC) colonic volumes, measured by MRI, in mL Data given: AUC for total colon Measurements at 0, 1, 2, 3, 4, 5, 6, 7, and 8 hours post-intervention
Time Frame: 0 - 8 hours
Measure: Mean (Standard Deviation); unit: ml*minutes
Arm/Group | Kiwifruit | Control
Number analyzed (Participants) | 14 | 14
ml*minutes | 283583 (59402) | 243182 (46682)

4. Secondary Outcome: Colonic Transit Time
Description: Transit of markers through gut as assessed by the weighted average position score (total score 0-7, calculated from a score of 0-7 of each of the 5 marker pills) at 24 h on MRI A lower score indicates faster transit.
Time Frame: 24hr
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Kiwifruit | Control
Number analyzed (Participants) | 14 | 14
Score on a scale | 0.8 [0 to 1.4] | 1.0 [0.5 to 3.1]

5. Secondary Outcome: Bowel Habit
Description: Assessment, via Diary, of bowel frequency Data given: stool frequency
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: stools per day
Arm/Group | Kiwifruit | Control
Number analyzed (Participants) | 14 | 14
stools per day | 1.46 (0.66) | 1.14 (0.46)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Kiwifruit | Control
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
This mechanistic study was limited by small sample size which was exacerbated by some participants' withdrawal from the study.

Did not control any other aspects of diet

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT03303417/Prot_SAP_ICF_000.pdf